CLINICAL TRIAL: NCT05557708
Title: Biodistribution of 68Ga Pentixafor in Patients With Small Cell Lung Carcinoma (SCLC)
Brief Title: A Safety Study of 212Pb-Pentixather Radioligand Therapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yusuf Menda (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Yusuf Menda, Professor and Director, Nuclear Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPORE Project 2; 1P50CA302572-01 (NIH)
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Carcinoid Tumor Lung; Neuroendocrine Tumor of the Lung; Carcinoma, Small-Cell Lung
Keywords: radioligand therapy; pentixather; Lead 203; Lead 212; alpha therapy; dosimetry
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 212-Lead Pentixather (Experimental): Single intravenous infusion of Pentixather radiolabeled with Lead-212. Administered activity to participant is calculated from bone marrow and renal radiation constraints.
  Treatment is administered in 2 cycles with 6 weeks between the cycles.
  Interventions: Drug: 212-Lead Pentixather; Diagnostic Test: 203-Lead Pentixather SPECT/CT

INTERVENTIONS:
Drug: 212-Lead Pentixather — Pentixather radiolabeled with 212-lead to target malignant cells with the CXCR4 ligand.
Diagnostic Test: 203-Lead Pentixather SPECT/CT — Pentixather radiolabeled with 203-Lead to identify the CXCR4 ligand on the malignant lesions for dosimetric analysis and treatment planning.

SUMMARY:
This is a first-in-human clinical trial evaluating the safety of an alpha-radiation treatment (Lead-212 labelled Pentixather) in patients who have been diagnosed with, and previously treated, for atypical carcinoid lesions of the lung.

DETAILED DESCRIPTION:
This is a study to determine what dose is acceptably safe for further testing.

In this study, participants are asked to:

* undergo SPECT/CT imaging with Lead-203 Pentixather (a radiotracer) to ensure the tumor lesions have the needed receptors
* undergo serial blood sampling for during and after the SPECT/CT scan for radiation and dosimetry calculations (to determine how much of the Lead-212 Pentixather to administer)
* receive up to 2 infusions of arginine & lysine as a kidney protectant
* receive up to 2 infusions of Lead-212 Pentixather, 6 weeks between each infusion
* undergo imaging at 3 months post treatment to determine disease response

ELIGIBILITY:
Inclusion Criteria:

* ability to provide independent consent
* adequate bone marrow function (platelet count ≥ 100,000; hemoglobin of ≥ 10 g/dL; neutrophil count ≥ 1,500 cells/mm3)
* adequate kidney function (creatinine clearance of ≥ 50 mL/min using the Cockcroft-Gault equation
* adequate liver function (serum bilirubin ≤ 3x the upper limit of normal, AST ≤ 5x the upper limit of normal, and ALT ≤ 5x the upper limit of normal)
* failed initial therapy or declined further therapy known to confer benefit
* have at least one lesion ≥ 2 cm that is positive for CXCR4 as demonstrated by Lead-203 Pentixather SPECT/CT

Exclusion Criteria:

* major surgery within 4 weeks of consent
* antoher investigational agent within 4 weeks of consent
* uncontrolled illness including, but not limited to, ongoing or active infection that would necessitate a delay in therapy or cause a hospital admission, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hepatic cirrhosis or severe impairment, or psychiatric illness/social situations that would limit compliance with study requirements.
* prior solid organ transplant
* cytotoxic or antineoplastic therapy within 21 days of consent (42 days for nitrosoureas)
* antibody therapy within the 21 days of consent
* allogenic bone marrow or stem cell transplant, or any stem cell infusion, within 84 days of consent
* pregnancy
* breastfeeding
* refusal to comply with birth control requirements during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine the recommended phase 2 dose of 212-Lead Pentixather | 3 months
  The recommended phase 2 dose is based on the number of dose limiting toxicities observed post-treatment.

SECONDARY OUTCOMES:
Determine the targeting of atypical pulmonary neuroendocrine tumor and/or neuroendocrine carcinoma lesions with 203-Lead Pentixather SPECT/CT | baseline
  The number of lesions identified with 203-Lead Pentixather SPECT/CT will compared to FDG PET/CT and diagnostic CT scans at baseline.
Determine tumor response | 3 months
  Tumor response will be assessed using the Response Evaluation Criteria in Solid Tumours (RECIST, v 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Menda, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data are obtained from protected health information. Only data from study participants who consented to data sharing will be shared.
  Data type:
  * patient demographics (age at consent, self-identified race ethnicity and gender, insurance status)
  * tumor response (RECIST measures, imaging DICOM)
  * adverse event logs indicating CTCAEv5 term and severity on a per-subject basis
  * dosimetric analysis of 203-Lead Pentixather scans
  * dose limiting toxicities: type and incidence
  * diagnostic analysis of 203-Lead Pentixather and FDG PET/CT (or CT) scans
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Protocol and ICF are made available upon request by email. All documents (Protocol, ICF, SAP, CSR, and analytic code) will be made available after primary objective is completed.
Access Criteria: A materials transfer agreement or data usage agreement (depending upon the legal department's preference) will need to be fully executed prior to sharing.

REFERENCES:
- [Background] Schottelius M, Osl T, Poschenrieder A, Hoffmann F, Beykan S, Hanscheid H, Schirbel A, Buck AK, Kropf S, Schwaiger M, Keller U, Lassmann M, Wester HJ. [177Lu]pentixather: Comprehensive Preclinical Characterization of a First CXCR4-directed Endoradiotherapeutic Agent. Theranostics. 2017 Jun 11;7(9):2350-2362. doi: 10.7150/thno.19119. eCollection 2017. PMID 28744319
- [Background] Buck AK, Serfling SE, Lindner T, Hanscheid H, Schirbel A, Hahner S, Fassnacht M, Einsele H, Werner RA. CXCR4-targeted theranostics in oncology. Eur J Nucl Med Mol Imaging. 2022 Oct;49(12):4133-4144. doi: 10.1007/s00259-022-05849-y. Epub 2022 Jun 8. PMID 35674738
- [Background] Serfling SE, Lapa C, Dreher N, Hartrampf PE, Rowe SP, Higuchi T, Schirbel A, Weich A, Hahner S, Fassnacht M, Buck AK, Werner RA. Impact of Tumor Burden on Normal Organ Distribution in Patients Imaged with CXCR4-Targeted [68Ga]Ga-PentixaFor PET/CT. Mol Imaging Biol. 2022 Aug;24(4):659-665. doi: 10.1007/s11307-022-01717-1. Epub 2022 Mar 21. PMID 35312939